CLINICAL TRIAL: NCT01348932
Title: The Relationship Between Single Nucleotide Polymorphisms of Chitinase 3-like 1 Gene,YKL-40 Serum Levels and Adult Asthma
Acronym: CHI3L1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Chen Chia-Hung, China Medical University Hospital
Other Study IDs: DMR100-IRB-008
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
Keywords: asthma; Chitinase 3-like 1 (CHI3L1); YKL-40; single nucleotide polymorphism(SNP); Real time PCR; gene
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The objective of this study was to investigate the relationship between single nucleotide polymorphism of chitinase 3-like 1 and human asthma. The association between CHI3L1 SNPs and the continuous outcomes were examined by real time PCR and gene sequencing analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Asthma: The relationship between single nucleotide polymorphisms of chitinase 3-like 1 gene, YKL-40 serum levels and adult asthma

SUMMARY:
The objective of this study was to investigate the relationship between single nucleotide polymorphism of chitinase 3-like 1 and human asthma.

DETAILED DESCRIPTION:
Chitinase 3-like 1 (CHI3L1) is a member of human chitinases family. According to previous studies in literatures, increased expression of CHI3L1 has been proven to be correlated with the presence of different diseases, including cancers, autoimmune diseases, and chronic inflammatory conditions. Elevated serum levels of YKL-40 are associated with increased disease severity, poorer prognosis and shorter survival for many other diseases. When monitored over time, increases in serum YKL-40 parallel with disease progression. It can serve as an measurable marker of changes in disease status.

There were indicated that chitinase 3-like 1 might be associated with some clinical diseases. The C-allele of the -131 C→G (rs4950928) polymorphism of CHI3L1 has been shown to associate with bronchial hyperresponsiveness and reduced lung function. It is suggesting that variations in CHI3L1 may influence risk of asthma.

The objective of this study was to investigate the relationship between single nucleotide polymorphism of chitinase 3-like 1 and human asthma. The association between CHI3L1 SNPs and the continuous outcomes were examined by real time PCR and gene sequencing analysis.

In Korean reports there was no significant associations between CHI3L1 SNPs and asthma were observed. On the other hand, there were association between CHI3L1 and asthma observed in the majority of Caucasian populations. However, similar research has not been conducted in Taiwan. In contrast to preliminary studies, the investigators predict the rs4950928 G allele, and not the C allele, was found to be associated with asthma. The g.-247C/T polymorphism in the CHI3L1 promoter region is associated with the risk of atopy.

ELIGIBILITY:
Inclusion Criteria:

* ages 20 to 60 years
* asthma patients
* atopy patients
* control (non-asthma and non-atopy)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Taiwan
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-06 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chia Hung, doctor, Study Director — Partners
Locations (1):
- China Medical University Hospital, 2 Yuh-Der Road, Taichung, Taiwan